CLINICAL TRIAL: NCT00963560
Title: A Randomized, Subject-masked Comparison of Visual Function After Bilateral Implantation of Presbyopia-correcting IOLs
Brief Title: Presbyopia-Correcting Intraocular Lenses (IOLs)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Diane Houtman, Director - Global Scientific Market Affairs Dept, Alcon Laboratories, Inc.
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: M09-008
Record Dates: First submitted 2009-08-19; First posted 2009-08-21 (Estimated); Results first posted 2011-08-09 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-07

CONDITIONS: Cataract
Keywords: ReSTOR +3
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- ReSTOR +3 (Experimental): Bilateral implantation of ReSTOR +3 Intraocular Lens (IOL)
  Interventions: Device: ReSTOR +3
- Crystalens HD (Active Comparator): Bilateral implantation of Crystalens HD Intraocular Lens (IOL)
  Interventions: Device: Crystalens HD
- Crystalens AO (Active Comparator): Bilateral implantation of Crystalens AO Intraocular Lens (IOL)
  Interventions: Device: Crystalens AO

INTERVENTIONS:
Device: ReSTOR +3 — Bilateral implantation of the AcrySof ReSTOR Aspheric +3 Model SN6AD1 Intraocular lens (IOL) for the treatment of cataract.
  Arms: ReSTOR +3
Device: Crystalens HD — Bilateral implantation of the Crystalens HD intraocular lens (IOL) for the treatment of cataract.
  Arms: Crystalens HD
Device: Crystalens AO — Bilateral implantation of the Crystalens AO intraocular lens (IOL) for the treatment of cataract.
  Arms: Crystalens AO

SUMMARY:
The purpose of this study is to prospectively evaluate postoperative visual and refractive parameters in a series of subjects bilaterally implanted with Presbyopia-Correcting Intraocular Lenses (IOLs).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with bilateral cataracts
* candidate for presbyopic lens

Exclusion Criteria:

* > 1 Diopter preoperative astigmatism by Keratometry readings
* pre-existing conditions that could skew the results

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2009-08; Primary Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center For Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Bilateral diagnosis of cataracts of subjects >21 years of age.
Pre-assignment Details: During the preoperative exam, subjects were examined to ensure they met the inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | ReSTOR +3 | Crystalens HD | Crystalens AO
Started | 47 | 44 | 41
Completed | 44 | 41 | 41
Not Completed | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ReSTOR +3 | Crystalens HD | Crystalens AO | Total
Number analyzed (Participants) | 47 | 44 | 41 | 132
Age Continuous [Mean (Standard Deviation); unit: years] | 63.4 (9.4) [41 to 81] | 64 (7.8) [50 to 79] | 65.3 (7.5) [50 to 81] | 64.23 (8.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 26 | 79
  Male | 19 | 19 | 15 | 53

OUTCOME MEASURES:

1. Primary Outcome: Best Corrected Visual Acuity
Description: Best corrected vision was tested at 4 meters (m), 60 centimeters (cm), 40cm and at preferred distance (distance chosen by each subject) with a standard ETDRS chart for distance and a hand held chart for near. Scores were calculated using logMAR values. LogMAR is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better visual acuity. Preferred distance for each study group was as follows: ReSTOR +3 = 38.7 +/- 6.8 cm, Crystalens HD = 49.9 +/- 9.8 cm, Crystalens AO = 53.1 +/- 9.8 cm.
Time Frame: 6 Months after surgery
Population: 2 ReSTOR +3 subjects and 1 Crystalens HD subject missed their final visits and were not included in this analysis.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR +3 | Crystalens HD | Crystalens AO
Number analyzed (Participants) | 42 | 40 | 41
logMAR
  4m (far) Distance | -0.075 (0.100) | -0.080 (0.103) | -0.081 (0.110)
  60cm (intermediate) Distance | 0.227 (0.119) | 0.176 (0.139) | 0.200 (0.154)
  40 cm (near) Distance | 0.057 (0.086) | 0.364 (0.183) | 0.420 (0.188)
  Preferred Distance | 0.055 (0.121) | 0.223 (0.146) | 0.222 (0.138)

ADVERSE EVENTS:
Time Frame: Day of surgery until visit 6 months following surgery.
Arm/Group | ReSTOR +3 | Crystalens HD | Crystalens AO
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/44 | 0/41
Other Adverse Events (participants affected / at risk) | 0/47 | 0/44 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data and discoveries arising out of the study, patentable or nonpatentable, shall be the sole property of Alcon Laboratories, Inc. Alcon reserves the right of prior review of any publication or presentation of information related to the study. Alcon may use these data now and in the future for presentation or publication at Alcon's discretion or for submission to government regulatory agencies.